CLINICAL TRIAL: NCT02842112
Title: Higher Percentage of CD34+ CD38- Cells Detected by Multiparameter Flow Cytometry From Leukapheresis Products Predicts Unsustained Complete Remission in Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0460
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; prognosis; stem cell harvest; autologous transplant; leukemia stem cell
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute | interventions — Leukapheresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CD34+ CD38-: A first cell population, which expressed the CD34 antigen and lacked CD38 (CD34+ CD38-), and often contained very few events requiring to be tightly clustered in a forward light scatter /side light scatter (FSC/ SSC) and CD45/SSC plot;
  Interventions: Other: PBSC mobilization and leukapheresis
- CD34+ CD38low: A second population characterized by expression of the CD34 antigen and by a low density of CD38 antigen (CD34+ CD38low)
  Interventions: Other: PBSC mobilization and leukapheresis
- CD34+ CD38+: A third population characterized by a large density of CD38 and CD34 antigens (CD34+ CD38+). Antigens were expressed as percent positively stained cells as well as intensity of the fluorescence signal quantified as mean fluorescence intensity (MFI) from CD34+ gated cells and from CD45low/SSC total immature cells
  Interventions: Other: PBSC mobilization and leukapheresis

INTERVENTIONS:
Other: PBSC mobilization and leukapheresis — Mobilization and harvest of autologous PBSCs was scheduled during the recovery phase after the consolidation course. Granulocyte colony stimulating factor (G-CSF) (150 µg/m2/day) was given by daily subcutaneous injection from day 20 of the chemotherapy course until completion of the blood stem cell collections. PBSC collections were performed on 1 - 5 consecutive days during the hematopoietic recovery phase, as soon as the leukocyte count exceeded 2x 109/L.
  Collections were performed after induction or after consolidation. In cases in which the minimum number of CD34+ cells was not collected, an additional mobilization was performed in steady state.
  Harvesting was performed using continuous flow blood cell separators. Cells were stored in liquid nitrogen until use, according to standard techniques.

SUMMARY:
Over recent decades, improvements have been made in the treatment of adult acute myeloid leukemia (AML). This has been mainly attributed to improvements in supportive therapy and to intensification of treatment strategies. The introduction of a post-induction myeloablative regimen followed by allogeneic stem cell transplant (SCT) has reduced the relapse rate in younger adults. However, this procedure is limited by the availability of human leukocyte antigen (HLA)-identical donors and conventional SCT preparative regimens according to patient age. In the absence of a compatible donor, myeloablative chemotherapy followed by autologous peripheral blood (PB) SCT remains one treatment strategy in adult patients with AML, allowing 35 - 50% long-term survivors. Despite several advantages of the CD34+ cell mobilization procedure, recent data have shown that relapse was higher and leukemia-free survival (LFS) shorter compared with bone marrow (BM) autografts. Higher doses of CD34+ peripheral blood stem cells (PBSCs) are collected to ensure engraftment and possibly reduce the incidence of treatment-related mortality (TRM). Although there is a threshold CD34+ cell dose below which engraftment is delayed in AML, the positive linear correlation of the number of CD34+ cells and kinetics of engraftment reaches a limit above which an increase in the number of progenitor cells does not provide any additional benefit. Relapse has been shown to be higher and survival shorter for those who receive the highest CD34+ PB doses. Although highly active against the leukemia bulk, intensive chemotherapy often spares the hardiest leukemia stem cells (LSCs) responsible for relapse. Detection of minimal residual disease (MRD) in autologous PBSC products may reflect inadequate in vivo purging, at least in part responsible for relapse. Although representing a heterogeneous cell population including both normal and leukemia cells, and despite that recent data have challenged the CD34+ CD38- phenotype of LSCs in AML, the CD34+ CD38- cell population generally remains considered enriched for LSCs.

In this setting, MRD remaining during morphological complete remission (CR) should be relatively enriched in CD34+ CD38- leukemia cells, and their persistence after CR achievement should correlate with disease recurrence. This was investigated in a cohort of 123 patients with AML following apheresis procedures after CR achievement. The investigators also studied the impact of the infused dose of subpopulations of CD34+ PB cells on the outcome of a subset of 71 patients who further underwent autologous PBSCT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* With a newly diagnosed de novo or secondary type AML (post myelodysplastic syndrome (MDS) or therapy-related AML)
* Patients achieving first CR after induction or salvage therapy

Exclusion Criteria:

* Patients with acute promyelocytic leukemia (APL)
* Concomitant uncontrolled infection, organ dysfunction or medical disease
* left ventricular ejection fraction (LVEF) < 45% as assessed by echocardiography

Ages: 25 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a newly diagnosed de novo or secondary type AML (post myelodysplastic syndrome MDS or therapy-related AML) and achieving first CR after induction or salvage therapy. Three populations of CD34+ cells were distinguished based on differential expression of the CD34 and CD38 antigens
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | During the study (1 year)
  EFS was defined from date of first apheresis to the date of relapse or death, or last contact with the patient in continuous complete remission

SECONDARY OUTCOMES:
Overall survival (OS) | During the study (1 year)
  OS was defined as the time from first apheresis to death or last patient contact. For patients effectively autografted, OS and EFS were calculated from the date of autologous SCT

CONTACTS AND LOCATIONS:
Overall Officials: Xavier THOMAS, MD-PhD, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud
Locations (1):
- Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, 165 Chemin du Grand Revoyet, Pierre-Bénite, France